CLINICAL TRIAL: NCT05978661
Title: A Single-Center Exploratory Study to Evaluate the Safety and Efficacy of FKC288 in Subjects With Relapsed or Refractory Systemic Light Chain (AL) Amyloidosis
Brief Title: FKC288 for Relapsed or Refractory Systemic Light Chain (AL) Amyloidosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-2301
Record Dates: First submitted 2023-05-07; First posted 2023-08-07 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Light Chain Amyloidosis
Keywords: AL Amyloidosis; BCMA/CD19-CAR-T cell
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: FKC288

INTERVENTIONS:
Drug: FKC288 — Administration of FKC288 Four dose groups of 0.1×10^6 CAR-T/kg, 0.3×10^6 CAR-T/kg, 1.0×10^6 CAR-T/kg, and 3.0×10^6 CAR-T/kg FKC288 are designed in this study. 3 to 6 subjects are expected to be enrolled in each dose group according to observed DLT.

SUMMARY:
This study is a single-center exploratory clinical trial. It is estimated that 6-12 subjects will be enrolled. The "BOIN" dose escalation design is adopted. The main purpose is to evaluate the safety of FKC288 in the treatment of subjects with relapsed or refractory AL amyloidosis and explore the recommended phase II dose of FKC288 in the treatment of patients with relapsed/refractory systemic Light Chain (AL) amyloidosis.

DETAILED DESCRIPTION:
A leukapheresis procedure will be performed to manufacture FKC288 chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of FKC288 at 0.1, 0.3, 1.0, or 3.0x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after FKC288 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must personally sign a written informed consent form approved by the ethics committee before the start of the study;
2. The subject's age is ≥18 years old and <70 years old;
3. The subject must be diagnosed with light chain amyloidosis by pathological examination, with at least one major organ involved (heart, kidney, or liver);
4. The subject with recurrent/refractory light chain amyloidosis that achieved no response with conventional treatment;
5. dFLC > 50mg/L;
6. Expected survival ≥ 12 weeks;
7. ECOG score ≤ 2 points;
8. Female subjects with fertility should agree to practice an effective method of contraception from the day of signing the ICF until 365 days after the infusion. An effective method of contraception is defined as abstinence or contraceptive methods with an annual failure rate of <1% specified in the plan.
9. Before enrollment, the subject must have appropriate organ function and meet all the following criteria:

1) Absolute neutrophil count ≥ 1.0×109/L (use of granulocyte colony-stimulating factor (G-CSF) support is allowed, but must be without supportive treatment within 7 days before the examination); 2) Platelet count ≥ 75×109/L (no transfusion support [including component transfusion] or treatments aimed at raising platelets such as thrombopoietin [TPO] should be received within 7 days before the examination); 3) Hemoglobin ≥ 9 g/dl (no transfusion support [including component transfusion] should be received within 7 days before the examination); 4) Bilirubin value ≤ 1.5× upper limit of normal (ULN) (except bile duct obstruction caused by tumor compression); 5) Creatinine clearance rate ≥ 40 ml/min; 6) ALT or AST ≤ 2.5× ULN (≤5 times the upper limit of normal in patients with liver involvement); 7) Echocardiography results indicate left ventricular ejection fraction ≥ 50% with no significant pericardial effusion; 8) NTproBNP < 1800pg/ml, TNT < 0.06ng/ml; 9) Stable coagulation function: INR ≤ 1.5, APTT ≤ 1.2× ULN (excluding tumor-related anticoagulant therapy); 10) >95% basic blood oxygen saturation in the natural indoor air environments.

Exclusion Criteria:

1. Subjects who have received any of the following treatments prior to enrollment: 1) Subjects who have received gene therapy before enrollment; 2) Subjects who have received live vaccines within 4 weeks prior to enrollment; 3) Subjects has received other interventional clinical research drugs within 12 weeks before apheresis.
2. Subjects with central metastasis or complete intestinal obstruction.
3. Subject with moderate or more severe hydrothorax and ascites which are hard to control by conventional treatment and require continuous catheter drainage.
4. With an active malignant tumor in the past 5 years, unless it is a curable tumor and has been obviously cured.
5. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and have abnormal peripheral blood HBV DNA test results (HBV DNA test abnormality is defined as HBV DNA quantitative detection is higher than the detection center's detection lower limit or higher than the detection center's normal reference range or HBV DNA qualitative detection is positive); hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; human immunodeficiency virus (HIV) antibody positive; the cytomegalovirus (CMV) DNA positive; syphilis testing RPR positive.
6. Presence of uncontrollable active infections (excluding <CTCAE grade 2 urinary and respiratory tract infections).
7. Severe cardiovascular diseases, including but not limited to unstable angina pectoris, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), and severe arrhythmias.
8. Subjects with hypertension that cannot be controlled by medication.
9. Toxicity reactions that have not been relieved to baseline or ≤ grade 1 (NCI-CTCAE version 5.0, except for hair loss and laboratory test abnormalities without clinical significance) from past treatments.
10. Major surgery within 2 weeks before enrollment, or has a surgery planned during the time the subject is expected to be infused with FKC288 or within 12 weeks after FKC288 infusion (except planned surgery under local anesthesia).
11. Subject who has a solid organ transplant.
12. Women who are pregnant or breastfeeding.
13. Subjects with previous central nervous system diseases (such as cerebral aneurysm, epilepsy, stroke, dementia, psychosis, etc.) or conscious disorders.
14. Other systemic diseases that the investigator judges as unstable, including but not limited to severe liver, kidney, or metabolic diseases that require medication.
15. Known life-threatening allergic reactions, hypersensitivity reactions, or intolerance to FKC288 cell preparations or their components.
16. Subjects judged by the investigator to have bleeding or severe thrombosis, or have inherited/acquired bleeding and severe thrombosis (including hemophilia, coagulation dysfunction, thrombocytopenia, splenomegaly, etc.), or are receiving thrombolysis or anticoagulation therapy.
17. Other situations deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with dose-limiting toxicity | Within 28 days after FKC288 injection infusion
  The number of participants with dose limiting toxicity in each dose group and the type of dose limiting toxicity that occurred.
The proportion of subjects with adverse events | Within 24 weeks after FKC288 injection infusion
  All adverse events were evaluated according to NCI-CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Proportion of subjects achieving hematologic response | Within 6 months after FKC288 injection infusion
  The proportion of subjects who achieve any type of hematologic response according to the 2023 National Comprehensive Cancer Network (NCCN) systemic light-chain amyloidosis guidelines within 6 months after receiving FKC288 infusion.
Proportion of subjects achieving organ response | Within 2 years after FKC288 injection infusion
  The proportion of subjects who achieve any type of organ response according to the 2023 National Comprehensive Cancer Network (NCCN) systemic light-chain amyloidosis guidelines within 2 years after receiving FKC288 infusion.
Progression-free survival (PFS) of all subjects | Within 2 years after FKC288 injection infusion
  Time from the first FKC288 infusion to the first assessment of disease progression/relapse or death from any cause.
Overall survival (OS) of all subjects | Within 2 years after FKC288 injection infusion
  Time from the first FKC288 infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xianghua Huang, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No